CLINICAL TRIAL: NCT06900192
Title: A Multicenter Phase 1 Study of Allogeneic Hematopoietic Cell Transplantation for Primary Progressive Multiple Sclerosis Using Orca-Q, an Engineered Donor Graft Derived From Mobilized Peripheral Blood
Brief Title: A Study of Allogeneic Hematopoietic Cell Transplantation for Primary Progressive Multiple Sclerosis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Orca Biosystems, Inc. (Industry)
Responsible Party: Principal Investigator, Everett Meyer, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 75412
Record Dates: First submitted 2025-02-03; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Primary Progressive Multiple Sclerosis; Multiple Sclerosis; Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Secondary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Busulfan; fludarabine; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Orca-Q Graft with lymphodepleting conditioning regimen (Experimental): Donor Orca-Q stem cell graft
  Interventions: Biological: Orca-Q; Drug: myeloablative regimen

INTERVENTIONS:
Biological: Orca-Q — Allogeneic (donor) stem cell graft
Drug: myeloablative regimen — Myeloablative regimen of busulfan, fludarabine, and thiotepa.
  Other Names: busulfan; fludarabine; thiotepa

SUMMARY:
A study of alloHCT with Orca-Q for the treatment of primary progressive multiple sclerosis (MS).

DETAILED DESCRIPTION:
This study will evaluate alloHCT with Orca-Q, an allogeneic hematopoietic graft isolated from a donor's hematopoietic cells for the treatment of primary progressive MS.

ELIGIBILITY:
Inclusion Criteria (Recipient):

1. Participants aged ≥18 and ≤65 years with primary progressive multiple sclerosis
2. A diagnosis of PPMS by 2017 McDonald criteria and 2013 clinical course revision102
3. CSF with elevated IgG index or 2 or more oligoclonal bands
4. EDSS (see Appendix 9) between 2.0 and 5.5 inclusive
5. Based on review of the clinical records, there must be a deterioration in the EDSS of at least 1 or more points over the previous 4 years (or less).
6. Eligibility criteria confirmed by the Eligibility Review Group (Appendix 10)
7. Recipients who have been treated with ocrelizumab, rituximab, ofatumumab, ublituximab, or alemtuzumab must undergo a washout period as described in Appendix 14 prior to their planned day 0.
8. Recipients must be willing to undergo mobilized autologous peripheral blood stem cell collection to create a cryopreserved rescue product prior to alloHCT.
9. Ability to undergo MRI without general anesthesia
10. Ability to undergo all tests and procedures in the study
11. Patients who are not vaccinated for COVID-19 must have no symptoms of COVID-19 and have negative testing for COVID-19. For other vaccine-preventable illnesses, it is recommended that patients are current on their vaccination schedule.

Exclusion Criteria:

1. History of Progressive Multifocal Leukoencephalopathy
2. Organ dysfunction or disease that would jeopardize survival after hematopoietic cell transplantation, including but not limited to the following:

   1. Renal insufficiency as defined by an estimated GFR <60 mL/minute
   2. Cardiac dysfunction as defined by symptomatic coronary artery disease, congestive heart failure, valvular heart disease, cardiomyopathy, uncontrolled arrhythmia(s), or left ventricular ejection fraction <50%. Participants with a history of these conditions may enroll if they are demonstrated to have optimal cardiac function (as defined by echocardiography or multi-gated acquisition scan)
   3. Pulmonary dysfunction that poses a risk of mortality after transplant, defined as pre-transplant pulmonary function testing demonstrating a FEV1 <70% expected and/or a DLCOadj <70% expected.
   4. Necroinflammatory or fibrotic liver disease with evidence of liver dysfunction, including but not limited to jaundice, hepatic encephalopathy, or portal hypertension
   5. Marrow dysfunction that poses a risk of peri-transplant mortality, defined as an absolute neutrophil count (<1000/mm3) below the lower limit of normal, or a platelet count below 50,000/mm3.
   6. Poorly controlled hypertension despite appropriate therapy, defined as a diastolic blood pressure greater than 90 mm Hg while on therapy.
   7. Poorly controlled diabetes mellitus, defined as HgbA1c ≥ 6.5% despite therapy or recurrent hypoglycemia while on therapy.
   8. Extreme protein-calorie malnutrition defined by Body Mass Index <18 and unintentional weight loss (3 kg in the last month or 6 kg in the last 6 months.)
3. History of smoking either tobacco or other herbal products in the last 3 months.
4. Planned pharmaceutical in vivo or ex vivo T cell depletion (TCD), eg, cladribine, or peritransplant antithymocyte globulin (ATG). For participants who have previously been exposed to a TCD agent, a 5-half-life washout of the agent must occur prior to planned day 0 (day 0 is defined as the day of infusion Orca-Q Prime). The washout period for alemtuzumab is listed in Appendix 14.
5. HIV seropositive.
6. HBV serology results indicating chronic HBV infection per https://www.cdc.gov/hepatitis/hbv/interpretationOfHepBSerologicResults.htm, unless HBV PCR negative. HBV seropositive participants should be on antiviral therapy after transplant.
7. HCV seropositive, unless PCR negative and having undergone 'curative' antiviral therapy.
8. Participant has active uncontrolled infection
9. Participant has demonstrated lack of compliance with prior medical care
10. Participants with known active malignancy. It is recommended that patients are current on cancer screening tests for their age and family history as per the NCCN [The National Comprehensive Cancer Network®] Guidelines. Screening should be performed, if indicated, per NCCN guidelines prior to study treatment.
11. Participants whose life expectancy is severely limited by illness other than multiple sclerosis
12. Females who are pregnant or breast feeding.
13. Medical or psychiatric conditions that compromise ability to give informed consent or to comply with treatment protocol
14. Inability to undergo an MRI scan
15. Currently receiving treatment with investigational agents
16. Positive for JC virus DNA in the CSF or blood during screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Severe acute Graft-versus-Host-Disease-free survival | 365 days after infusion
  Alive without a history of moderate to severe aGVHD

SECONDARY OUTCOMES:
Evaluate treatment response | Measurements will be taken at 9 and 12 months after infusion
  Neurologically stable. Assessment of neurological function will be measured by employing the expanded disability status scale (EDSS)
Evaluate safety of treatment | Measured from time of enrollment to end of study participation (from date of consent to month 12).
  Regimen-related toxicity, incidence and severity of GVHD, primary and secondary graft failure

IPD SHARING:
Plan to Share IPD: No